CLINICAL TRIAL: NCT01016730
Title: Single-Arm, Dose-Finding Pilot Trial of Single-Agent Bortezomib in Patients With Relapsed/Refractory AIDS-Associated Kaposi Sarcoma With Correlative Assessments of KSHV and HIV
Brief Title: Bortezomib in Treating Patients With Relapsed or Refractory AIDS-Related Kaposi Sarcoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2012-03170; NCI-2012-03170 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CDR0000659554; AMC-063 (Other: AIDS Malignancy Consortium); AMC-063 (Other: CTEP); U01CA121947 (NIH); UM1CA121947 (NIH)
Record Dates: First submitted 2009-11-18; First posted 2009-11-19 (Estimated); Last update posted 2018-02-20 (Actual); Status verified 2018-02

CONDITIONS: AIDS-Related Kaposi Sarcoma; HIV Infection; Recurrent Kaposi Sarcoma
MeSH Terms: conditions — AIDS-related Kaposi sarcoma; HIV Infections; Sarcoma, Kaposi | interventions — Bortezomib

ARMS (1):
- Treatment (bortezomib) (Experimental): Patients receive bortezomib IV on days 1, 8, and 15. Treatment repeats every 28 days for up to 8 courses in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Bortezomib; Other: Laboratory Biomarker Analysis; Other: Questionnaire Administration

INTERVENTIONS:
Drug: Bortezomib — Given IV
  Other Names: [(1R)-3-Methyl-1-[[(2S)-1-oxo-3-phenyl-2-[(pyrazinylcarbonyl)amino]propyl]amino]butyl]boronic Acid; LDP 341; MLN341; PS-341; PS341; Velcade
Other: Laboratory Biomarker Analysis — Correlative studies
Other: Questionnaire Administration — Ancillary studies

SUMMARY:
This pilot, phase I trial studies the side effects and best dose of bortezomib in treating patients with acquired immune deficiency syndrome (AIDS)-related Kaposi sarcoma that has come back or has not responded to treatment. Bortezomib may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Estimate the maximum tolerated dose (MTD) of single agent bortezomib in subjects with AIDS-related Kaposi sarcoma (KS).

SECONDARY OBJECTIVES:

I. Evaluate the clinical response of KS tumors to bortezomib. II. Evaluate the impact of bortezomib on human immunodeficiency virus (HIV) plasma viral loads and peripheral blood mononuclear cells (PBMC) apolipoprotein B messenger ribonucleic acid (mRNA) editing enzyme, catalytic polypeptide-like 3G (APOBEC3G) levels.

III. Determine the impact of bortezomib on Kaposi's sarcoma-associated herpesvirus (KSHV).

IV. Assess bortezomib effects on KSHV copy number in PBMC and plasma and whether changes in viral copy number measured in PBMC and plasma are associated with clinical response of KS tumors.

V. Monitor KSHV gene expression in KS biopsy specimens and PBMC pre- and post-bortezomib and assess whether changes in viral gene expression (i.e., to a lytic pattern) in tumor biopsy are associated with clinical response.

VI. Assess whether changes in viral copy number in PBMC and plasma occur in concert with or independently of changes in viral antigen expression in tumor biopsy specimens.

VII. Assess effects of bortezomib on proteins relevant to KS tumor survival and proliferation (i.e., P53, von Hippel-Lindau [VHL], p27, hypoxia-inducible factor 1 [HIF1]-alpha) as well as levels of nuclear factor-kappaB (NFkappaB) gene target mRNAs in tumor biopsies.

OUTLINE: This is a dose-escalation study.

Patients receive bortezomib intravenously (IV) on days 1, 8, and 15. Treatment repeats every 28 days for up to 8 courses in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up at 4 weeks and then every 3 months for up to 1 year.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients with cutaneous AIDS-related biopsy-proven KS relapsed after or refractory to at least one other prior systemic therapy
* Patients must have cutaneous KS lesion(s) amenable to biopsy (either one lesion >= 12 mm or 3 >= 4 mm) in addition to at least 5 lesions measurable for assessment; all of these lesions must not have been previously radiated
* Must have been on stable anti-retroviral therapy for at least 12 weeks with a principal investigator (PI)-based or non-nucleoside reverse-transcriptase inhibitor (NNRTI)-based regimen of at least three drugs, with no intention to change the regimen for the duration of the study; patients who have a high likelihood of better HIV management with a new antiretroviral regimen should defer enrollment until the changes are in place and the new highly active antiretroviral therapy (HAART) regimen meets the 12 week criteria
* Serologic documentation of HIV infection at any time prior to study entry, as evidenced by positive enzyme-linked immunosorbent assay (ELISA), positive western blot, or other Food and Drug Administration (FDA)-approved licensed HIV test, or a detectable blood level of HIV RNA
* Women of child-bearing potential must have a negative pregnancy test within 72 hours before initiation of study drug dosing; post-menopausal women must be amenorrheic for at least 12 months to be considered of non-childbearing potential; male and female subjects of reproductive potential must agree to employ an effective barrier method of birth control throughout the study and for up to 3 months following discontinuation of study drug; (Note: a woman of childbearing potential is one who is biologically capable of becoming pregnant; this includes women who are using contraceptives or whose sexual partners are either sterile or using contraceptives)
* Absolute neutrophil count (ANC) >= 1,000/mm^3; subjects may be receiving growth factor support to meet these criteria
* Hemoglobin >= 8.0 gm/dL; subjects may be receiving growth factor support to meet these criteria
* Platelets >= 100,000/mm^3
* Total bilirubin =< 1.5 mg/dL; if the elevated bilirubin is felt to be secondary to indinavir or atazanavir therapy, then subjects will be allowed on protocol without any limit on the total bilirubin if the direct bilirubin is normal
* Aspartate aminotransferase (AST) (serum glutamic oxaloacetic transaminase [SGOT]) and alanine aminotransferase (ALT) (serum glutamate pyruvate transaminase [SGPT]) =< 2.5 x institutional upper limit of normal (ULN)
* Serum creatinine =< institutional ULN or creatinine clearance >= 50 mL/min/1.73 m^2 for subjects with creatinine levels above institutional ULN
* Pre-existing grade 3 or 4 peripheral neuropathy

Exclusion Criteria:

* KS that is improving in the 4 weeks prior to enrollment
* Symptomatic visceral KS (oral and lymph node involvement is eligible)
* Symptomatic pulmonary KS; asymptomatic pulmonary KS that is not limiting activities of daily living is allowable
* Eastern Cooperative Oncology Group (ECOG) performance status greater than 2
* Expected survival < 3 months with standard KS treatments (i.e., radiation, paclitaxel)
* Concurrent active opportunistic infection (OI)
* Herpes zoster (shingles) outbreak within the last 6 months or inability to take herpes zoster prophylaxis
* Patient is =< 5 years free of another primary malignancy except if the other primary malignancy is neither currently clinically significant nor requiring active intervention, or if the other primary malignancy is a localized squamous or basal cell skin cancer or cervical/anal carcinoma in situ
* Acute treatment for an infection or other serious medical illness within 14 days prior to study entry
* Patients may not have had anti-neoplastic treatment for Kaposi sarcoma (including chemotherapy, radiation therapy, biological therapy, or investigational therapy) within 4 weeks (6 weeks for nitrosourea or mitomycin-C) of study treatment
* Prior treatment with bortezomib or other investigational proteasome inhibitors
* Previous local therapy of any KS indicator lesion within 60 days, unless the lesion has clearly progressed with enlargement since the local therapy
* Use of any investigational drug or treatment within 4 weeks prior to randomization
* Physical or psychiatric conditions that in the estimation of the investigator place the patient at high risk of toxicity or non-compliance
* Hypersensitivity to boron
* Subjects with grade III/IV cardiac disease as defined by the New York Heart Association criteria. (e.g., congestive heart failure, myocardial infarction within 6 months of study)
* Subject has an acute or known chronic liver disease (e.g., chronic active hepatitis, cirrhosis); subjects with known hepatitis B or C infection may be enrolled if they have either documentation of no or minimal fibrosis on liver biopsy or undetectable hepatitis virus on polymerase chain reaction (PCR)
* Systemic corticosteroid treatment, other than replacement doses
* Female subjects who are pregnant or breast-feeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2010-01-22 (Actual); Primary Completion 2015-01-07 (Actual); Study Completion 2015-01-07 (Actual)

PRIMARY OUTCOMES:
MTD based on the National Cancer Institute Common Terminology Criteria for Adverse Events version 4.0 | 56 days
  MTD is defined as the highest assigned dose at which < 2 patients (out of 6) experience dose-limiting toxicity. Adverse events will be summarized by type, timing, and severity grade.

SECONDARY OUTCOMES:
Change in lytic gene expression | Baseline to 1 year
  The association between change in lytic gene expression with clinical response of KS tumors will be investigated with exact logistic regression. Hierarchical clustering will be used to explore if gene expression patterns differ according to clinical response.
Changes in bortezomib in KSHV copy number in PBMC and plasma | Baseline to 1 year
  Analyzed using the Wilcoxon signed rank test. The association between change in KSHV copy number with clinical response of KS tumors will be investigated with exact logistic regression.
Changes in levels of tumor survival, proliferation proteins, and NFKappaB gene target mRNA levels | Baseline to 1 year
  Analyzed using the Wilcoxon signed rank test.
Changes in viral antigen expression in biopsy specimens | Baseline to 1 year
  Spearman's rank correlations will be calculated to examine whether the changes in KSHV viral copy number in PBMC and plasma occur in concert or independently with changes in viral antigen expression in biopsy specimens collected at baseline, day 2 and treatment discontinuation.
Clinical KS response rates based on the Response Evaluation Criteria in Solid Tumors | Up to 1 year
  Exact binomial 95% confidence intervals will be computed. Descriptive statistics will also be presented for complete and partial response rates.

CONTACTS AND LOCATIONS:
Overall Officials: Erin Reid, Principal Investigator — AIDS Malignancy Consortium
Locations (9):
- United States (9):
  - UC San Diego Moores Cancer Center, La Jolla, California
  - UCLA Center for Clinical AIDS Research and Education, Los Angeles, California
  - UCLA / Jonsson Comprehensive Cancer Center, Los Angeles, California
  - University of California San Diego, San Diego, California
  - Johns Hopkins University/Sidney Kimmel Cancer Center, Baltimore, Maryland
  - Boston Medical Center, Boston, Massachusetts
  - Memorial Sloan Kettering-Rockefeller Outpatient Pavilion, New York, New York
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - Virginia Mason Medical Center, Seattle, Washington